CLINICAL TRIAL: NCT01156974
Title: Care Guides: Can Trained Laypersons Help Manage Chronic Disease? A Randomized Trial.
Brief Title: Care Guides in the Primary Care Office (Phase II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3096-1E
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Diabetes; Hypertension; Congestive Heart Failure
Keywords: care management; chronic disease; outpatient
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Heart Failure; Chronic Disease | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- care guide (Experimental): patients receive education about care goals and work with a care guide to achieve goals
  Interventions: Behavioral: education and care guide
- no care guide (Active Comparator): patients receive education about care goals and usual care to achieve goals
  Interventions: Behavioral: education only

INTERVENTIONS:
Behavioral: education and care guide — Patients receive education about care goals, and in-person and telephone counseling of unspecified frequency over one year to achieve goals
  Other Names: Active care management
  Arms: care guide
Behavioral: education only — patients receive education about care goals
  Arms: no care guide

SUMMARY:
Trained lay persons ("care guides") working with chronic disease patients and their providers can help outpatients with diabetes, hypertension, and congestive heart failure achieve standard clinical care goals

DETAILED DESCRIPTION:
In a randomized parallel group multi-site trial looking at achievement of standard recommended treatment goals at baseline and one year later by 2135 patients with diabetes, hypertension, and congestive heart failure, we tested the hypothesis that adding a lay person with brief training to usual care would improve clinical outcomes. These "care guides" were culturally matched to patients served, similar to community health workers, but were located in 6 diverse primary care health clinics where they could meet patients face-to-face. They were asked to assist communication in both directions between providers and patients, taking advantage of their status as non-authority figures. They were given two weeks' training about these diseases and behavior change theory. This intervention was designed to be low cost, easy to implement, and to integrate into rather than change clinic work flow.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-79
* diagnoses of diabetes, hypertension, and/or congestive heart failure

Exclusion Criteria:

* pregnant
* unable to understand randomization process

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2135 (Actual)
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
change in number of care goals met | one year
  Predetermined care goals as recommended by national authorities such as American Diabetes Association, American Heart Association, JNC-7.

SECONDARY OUTCOMES:
Kinds of patients who benefit from working with a care guide | one year
  demographic, clinical, and attitudinal characteristics of patients who benefit

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Adair, MD, Principal Investigator — Allina Health System
Locations (1):
- Allina Hospitals and Clinics, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Adair R, Christianson J, Wholey DR, White K, Town R, Lee S, Britt H, Lund P, Lukasewycz A, Elumba D. Care guides: employing nonclinical laypersons to help primary care teams manage chronic disease. J Ambul Care Manage. 2012 Jan-Mar;35(1):27-37. doi: 10.1097/JAC.0b013e31823b0fbe. PMID 22156953
- [Result] Adair R, Wholey DR, Christianson J, White KM, Britt H, Lee S. Improving chronic disease care by adding laypersons to the primary care team: a parallel randomized trial. Ann Intern Med. 2013 Aug 6;159(3):176-84. doi: 10.7326/0003-4819-159-3-201308060-00007. PMID 23922063
- [Result] Wholey DR, White KM, Adair R, Christianson JB, Lee S, Elumba D. Care guides: an examination of occupational conflict and role relationships in primary care. Health Care Manage Rev. 2013 Oct-Dec;38(4):272-83. doi: 10.1097/HMR.0b013e31825f3df9. PMID 22728580